CLINICAL TRIAL: NCT00579930
Title: Cytogenetic and Molecular Genetic Studies in Bone Sarcomas
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 93-141
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer
Keywords: Bone; Soft Tissue
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor Tissue

SUMMARY:
To establish a serial ascertainement of specimens from patients with bone sarcomas to be used in ongoing cytogenetic and molecular genetic analyses. These data will be integrated and correlated with the established Orthopaedic Service clinical database.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing diagnostic biopsy or resection of their primary or metastatic bone sarcoma for therapeutic purposes.
* The specimen must be large enough to allow routine pathological analysis, with the specimen for research excised from residual tissue that would otherwise be discarded.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 1993-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To establish a serial ascertainement of specimens from patients with bone sarcomas to be used in ongoing cytogenetic and molecular genetic analyses. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ladanyi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org